CLINICAL TRIAL: NCT03916393
Title: A SINGLE BLIND, RANDOMIZED, CROSS-OVER STUDY IN HEALTHY ADULT PARTICIPANTS TO INVESTIGATE THE PALATABILITY OF ORAL FORMULATIONS OF PF-06651600 FOR PEDIATRIC USE
Brief Title: PF-06651600 Taste Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: B7981021; 2019-000108-13 (EudraCT Number)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Healthy Participants
Keywords: PF-06651600; Palatability; Bitrex; Taste Study
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PF-06651600 Treatment A (Experimental): Active pharmaceutical ingredient (API)solution in water
  Interventions: Drug: PF-06651600 20 mg
- PF-06651600 Treatment B (Experimental): API in sweetened solution
  Interventions: Drug: PF-06651600 20 mg
- PF-06651600 Treatment C (Experimental): API blend suspension in water
  Interventions: Drug: PF-06651600 20 mg
- PF-06651600 Treatment D (Experimental): API blend suspension in apple sauce
  Interventions: Drug: PF-06651600 20 mg
- Bitrex (Registered) Treatment E (Other): Positive control for bitterness
  Interventions: Other: Bitrex solution

INTERVENTIONS:
Drug: PF-06651600 20 mg — PF-06651600 in four (4) different oral formulations will be administered in different periods.
  Arms: PF-06651600 Treatment A; PF-06651600 Treatment B; PF-06651600 Treatment C; PF-06651600 Treatment D
Other: Bitrex solution — Bitrex solution at 0.5 ppm will be included in the treatment sequence together with the four PF-06651600 formulations.
  Arms: Bitrex (Registered) Treatment E

SUMMARY:
This is a single-blind, randomized, five (5)-period, cross-over study in healthy adult participants. A group of approximately 10 participants will assess the sensory attributes (taste and palatability) of 4 different formulations of an investigational product (PF-06651600 active pharmaceutical ingredient) and Bitrex (Registered) positive control in a specified sequence in 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations and other study procedures.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease Infection with Hepatitis B, C or HIV
* Participants with conditions that affect their ability to taste
* Participants who currently smoke

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting overall liking of drug formulation | Baseline through 20 minutes post dose
  Overall liking assesses the degree that a participant likes a drug formulation based on sensory attributes experienced by the participant after tasting a product. It is scored based on a measurement of taste questionnaire.
Percentage of subjects reporting overall liking of drug formulation | Baseline through 20 minutes post dose
  Overall liking assesses the degree that a participant likes a drug formulation based on sensory attributes experienced by the participant after tasting a product. It is scored based on a measurement of taste questionnaire.
Number of subjects reporting saltiness of drug formulation | Baseline through 20 minutes post dose
  Saltiness assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire
Percentage of subjects reporting saltiness of drug formulation | Baseline through 20 minutes post dose
  Saltiness assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire
Number of subjects reporting bitterness of drug formulation | Baseline through 20 minutes post dose
  Bitterness assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire
Percentage of subjects reporting bitterness of drug formulation | Baseline through 20 minutes post dose
  Bitterness assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire
Number of subjects reporting mouth feel of drug formulation | Baseline through 20 minutes post dose
  Mouth feel assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire
Percentage of subjects reporting mouth feel of drug formulation | Baseline through 20 minutes post dose
  Mouth feel assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire
Number of subjects reporting sourness of drug formulation | Baseline through 20 minutes post dose
  Sourness assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire
Percentage of subjects reporting sourness of drug formulation | Baseline through 20 minutes post dose
  Sourness assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire
Number of subjects reporting tongue/mouth burn from drug formulation | Baseline through 20 minutes post dose
  Tongue/mouth burn assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire
Percentage of subjects reporting tongue/mouth burn from drug formulation | Baseline through 20 minutes post dose
  Tongue/mouth burn assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire
Number of subjects reporting formulation preference | Baseline through 20 minutes post dose
  Formulation preference assesses the degree that a participant prefers a drug formulation based on sensory attributes experienced by the participant after tasting a product. It is scored based on a measurement of taste questionnaire.
Percentage of subjects reporting formulation preference | Baseline through 20 minutes post dose
  Formulation preference assesses the degree that a participant prefers a drug formulation based on sensory attributes experienced by the participant after tasting a product. It is scored based on a measurement of taste questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Be-bru, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7981021&StudyName=A+SINGLE+BLIND%2C+RANDOMIZED%2C+CROSS-OVER+STUDY+IN+HEALTHY+ADULT+PARTICIPANTS+TO+INVESTIGATE+THE+PALATABILITY+OF+ORAL+FORMULATIONS+OF+PF-06651600+FOR+PEDIATRIC+USE